CLINICAL TRIAL: NCT00246077
Title: Quality of Life of Children With Sickle Cell Disease Who Are Receiving Chronic Transfusion Therapy With a Lifeport Device
Brief Title: Quality of Life of Children With Sickle Cell Disease Who Are Getting Chronic Transfusions With a Lifeport
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: CMH 05 07-098E
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2005-11

CONDITIONS: Anemia, Sickle Cell
Keywords: chronic transfusion therapy; quality of life
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study is being done to see what impact having a Lifeport device has on quality of life for children with sickle cell who are getting chronic transfusions, from the child's perspective.

DETAILED DESCRIPTION:
There is a paucity of research that focuses specifically on quality of life (QoL) among patients with sickle cell. This study aims to explore the QoL of children who are receiving chronic transfusion therapy (CTT) using a Lifeport device, which allows them to undergo erythrocytapheresis, rather than standard transfusion therapy. Erythrocytapheresis is less time consuming and is associated with less iron overload than conventional transfusion therapy; however, little is known about the implications for the child's QoL. This study will explore QoL from the child's perspective.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of sickle cell disease between the ages of 8 & 18 years
* currently receiving chronic transfusion therapy via a Lifeport device
* Individuals have been utilizing the Lifeport for at least 6 months and no more than 18 months
* Individuals have received transfusions previously using conventional transfusion therapy (simple or exchange transfusions)
* Individuals have permission of parents (when applicable) and assent

Exclusion Criteria:

* Individuals who, in the opinion of the study staff, would suffer negative consequence, psychosocial trauma, or undue stress as a result of participation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5
Dates: Start 2005-10; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sarcone, RN, Study Director — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States